CLINICAL TRIAL: NCT04650711
Title: Immunohistochemical Staining of p16 for the Screening of Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CC-P16
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Cervical Cancer Screening; p16 Protein; Cytology; High-risk Human Papillomavirus; Diagnostic Accuracy; Histology; Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Intervention Model Description: All eligible participants as a cohort, accept P16INK4A testing, with cytology and/or hrHPV assay
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): All eligible participants as one group accept P16INK4A testing, with cytology and/or hrHPV assay.
  Interventions: Diagnostic Test: p16 protein expression

INTERVENTIONS:
Diagnostic Test: p16 protein expression — P16INK4A immunohistochemical staining is to be performed in residual cytology samples.
  Other Names: p16INK4A immunohistochemical staining

SUMMARY:
Cyclin kinase inhibitor P16INK4A has overexpression in cervical cancer, and hence becoming an alternative method for cervical cancer screening. This study is to investigate the clinical value of P16INK4A and high-risk human papillomavirus (hrHPV) detection of cervical intraepithelial neoplasia (CIN) 2 or more severe lesions (CIN2+). All eligible participants accept P16INK4A testing, with cytology and/or hrHPV assay. P16INK4A immunohistochemical staining is performed on the retained specimens of cytology. The primary endpoint is the diagnostic accuracy of P16INK4A compared with cytology and/or hrHPV status based on histology results. The accuracy analysis includes sensitivity, specificity, negative predictive value and positive predictive value.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Signed an approved informed consents
* With sufficient cytology sample for p16 testing
* With definite results of cytology and/or high-risk human papillomavirus and cervical histology

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-11-26 (Actual); Primary Completion 2020-11-26 (Estimated); Study Completion 2020-11-26 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of p16 protein expression | Two years
  Diagnostic accuracy of p16 protein expression for detecting cervical intraepithelial neoplasia (CIN) 2 or more severe lesions (CIN2+)

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China